CLINICAL TRIAL: NCT05982054
Title: Percutaneous Autologous Bone Marrow Cells With Core Decompression for Treating Avascular Hip Necrosis Under Local Anesthesia
Brief Title: Bone Marrow Cells With Core Decompression for AVN Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Global Stem Cell Center, Baghdad (Industry)
Responsible Party: Principal Investigator, abdulmajeed hammadi, GSCCBaghdad, Global Stem Cell Center, Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM protocol
Record Dates: First submitted 2023-07-18; First posted 2023-08-08 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Avascular Necrosis of the Femoral Head
Keywords: avascular necrosis of the femoral head; core decompression; bone marrow cells; local anesthesia
MeSH Terms: conditions — Femur Head Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bone marrow injection (Other): injection of autologous concentrated bone marrow cells under ultrasound and fluoroscopy guide after core decompression
  Interventions: Procedure: core decompression with local bone marrow mononuclear cells injection

INTERVENTIONS:
Procedure: core decompression with local bone marrow mononuclear cells injection — under local anesthesia ,anterior approach, with ultrasound and fluoroscopy guide

SUMMARY:
Avascular necrosis of the femoral head (AVN) is a progressive pathological process resulting from disruption of blood supply to the femoral head and elevation of intraosseous pressure. total hip arthroplasty is frequently the only durable option for pain relief and restoration of function. this is a single armed study to be done from July 2023 till January 2024, the total number of patients anticipated is 10, total joints treated around 20, The procedure includes core decompression with autologous bone marrow derived mononuclear cell injection inside the femoral head using local anesthesia ultrasound and fluoroscopy guided without drilling.

DETAILED DESCRIPTION:
Avascular necrosis of the femoral head (AVN) is a progressive pathological process resulting from disruption of blood supply to the femoral head and elevation of intraosseous pressure. Early stage AVN can be managed by various techniques, the results have been disappointing, total hip arthroplasty is frequently the only durable option for pain relief and restoration of function. This procedure is usually a high risk procedure under general anesthesia ,with The newer treatment modalities include using high stem cell concentration in the vicinity of the necrosed tissue with core decompression to prevent disease progression. this study is a single armed study to be done from July 2023 to January 2024, the total number of patients is 10, Etiology include corticosteroids use, systemic lupus erythematosus mostly related to steroid use in covid 19 epidemic,. The age of the patients range from 25-55 years. The procedure includes core decompression with autologous bone marrow derived mononuclear cell injection inside the femoral head using local anesthesia ultrasound and fluoroscopy guided without drilling.

ELIGIBILITY:
Inclusion Criteria:

1. Avascular hip necrosis irrespective Of stage.
2. age from 25-55 years. -

Exclusion Criteria:

1. history of bleeding tendency.
2. history of malignant disease.
3. critically ill patient. -

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
clinical improvement | 6 months
  change in Harris Hip Score which include 3 parameters 1-pain, 2-range of motion,3-function. maximum 100 which is excellent while 0 is bad.

SECONDARY OUTCOMES:
disease progression | around 6 months from starting recruitment
  percentage of patients who have clinical progress using Harris Hip Score which include 3 parameters 1-pain, 2-range of motion,3-function. maximum 100 which is excellent while 0 is bad or radiological proof of disease progression by Mitchell classification which is used to stage osteonecrosis of the femoral head and is based on MRI signal characteristics within the center of the lesion and classified into four stages with stage A representing early disease and stage D representing late disease.

CONTACTS AND LOCATIONS:
Overall Officials: abdulmajeed a hammadi, MD, Principal Investigator — clinical stem cell studies
Locations (1):
- Ministry of Health, Baghdad, Iraq